CLINICAL TRIAL: NCT00985803
Title: Comparison of Cardiovascular Training Versus Resistance Training In Patients With Systemic Lupus Erythematosus: Controlled Randomized Clinical Trial
Brief Title: Physical Activity in Patients With Systemic Lupus Erythematosus
Acronym: LESPA
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Marcelo Ismael Abrahão, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAbrahao
Record Dates: First submitted 2009-09-26; First posted 2009-09-28 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Activity Physical; Activity Disease,trials randomized
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group Control (No Intervention)
- Endurance (Experimental)
  Interventions: Other: Physical Activity: Endurance exercise training (ET)
- Cardiovascular (Experimental)
  Interventions: Other: Physical Activity: Cardio training (CT)

INTERVENTIONS:
Other: Physical Activity: Cardio training (CT) — The experimental group of resistance training will carry out the training with 8 kinds of training session with 12 reps with that load will vary according to the 1 RM test.
  The composition of the training session is 10 minutes of heating and stretching, 40 minutes of cardiovascular training and 10 minutes of cooling.
  Arms: Cardiovascular
Other: Physical Activity: Endurance exercise training (ET) — The experimental group of resistance training will carry out the training with 8 kinds of training session with 12 reps with that load will vary according to the 1 RM test.
  The composition of the training session is 10 minutes of heating and stretching, 40 minutes of cardiovascular training and 10 minutes of cooling.
  Arms: Endurance

SUMMARY:
The purpose of this study is to check the improvement in quality of life in patients with systemic lupus incorporated into a routine of physical activity.

Randomized controlled blinded trial, 63 patients aged 42.9 ± 14.4 and diagnosis of systemic lupus erythematosus (SLE) according to the criteria of the College American Rheumatology, 1997. After randomization patients were allocated into 3 groups, control group (CG) (n = 21), training cardiovascular (CT) (n = 20), resistance training (RT) (n = 22), performing 12 weeks of intervention with a frequency of three times weeks and were evaluated at two different times (T0 and T12). As primary outcome quality of life was assessed by the inventory Generic Assessment of quality of life by the Medical Outcomes Study 36 -- Healthy ItemShort Form Survey (SF36) and as secondary outcomes functional capacity evaluation of pain symptoms (visual scale analogue pain [VAS]), intensity of symptoms of depression (Beck Depression Inventory [BDI]), index of disease activity (Systemic Lupus Disease Activity Inventory Erythmatodud [SLEDAI]), capacity aerobic (walking test of 12 minutes [T12]), subjective perception effort (subjective scale of Borg [Borg]), limb muscle strength lower (analog dynamometer [strength]), electrical activity member lower (surface electromyography [EMG]), amount of products (inventory amount of Medicines).

DETAILED DESCRIPTION:
Will be selected 60 patients of both genders aged between 18 -55 years, with make the diagnosis of SLE by the criteria of the Americam College of Rheumatology revised in 1997 and that are not physically active.

After screening, patients will read and sign the informed consent form. The study will be submitted to the ethics committee of the Federal University of São Paulo / Escola Paulista de Medicina.

Randomization will be done by a secretary using a computer program specifically for this purpose, where the groups will be divided into intervention and control. The random allocation will be maintained using opaque sealed envelopes, which will open at the time of intervention.

Control group will not perform any type of training. Since the experimental group will be divided into two groups, cardio training (CT) and endurance exercise training (ET).

Evaluation will be conducted at the beginning and end of 12 weeks by two raters blind (who will not know to which groups, individuals were allocated) that will use the following tools:

* Outcomes
* Assessment of pain
* Assessment of pain before and after training, the visual analog scale of pain, ranging from 0 (zero) no pain and 10 cm (ten) 14 unbearable pain

Evaluation of the depression:

Evaluation of the depression at the beginning and end of the proposed training, inventory Beck Depression Inventory. (BDI). This inventory of multiple choice will be used to measure the severity of depression. These include symptoms of depression, irritability, cognitive impairment, guilt, feelings of being punished, physical symptoms such as fatigue, weight loss, lack of interest in sex.

Assessment of quality of life:

Generic Assessment of quality of life by the SF 36 (Short From 36), beginning and end of the proposed treatment. Validated in Portuguese in 1999 (Ciconelli et al, 1999). It consists of eight domains (physical functioning, limitation in physical appearance, bodily pain, general health, vitality, social, emotional, and mental health ranging from 0 (zero) to 100 (one hundred), and the higher the note is better quality of life.

Activity disease:

Activity Level by Systemic Lupus Erythematosus Disease Activity Inventory (SLEDAI) at the beginning and end of the proposed treatment.

Aerobic Capacity:

Cooper test of walking and / or running in 12 minutes. Only for the experimental group of aerobic training, aiming to prescribe the training range cardiovascular.O test aims to measure the aerobic capacity of subjects. The test results will be classified as "VERY GOOD", "GOOD", "MIDDLE", "BAD", "very poor", which will be based on distance traveled, age and sex of the individual being evaluated.

Muscle strength:

Evaluation of muscle strength through a load cell placed in a leg extension to 60 degrees of extension.

Activity Muscle:

Assessment of quadriceps muscle activation using electromyography

The experimental group of cardiovascular training will hold a training still between 55% to 65% of maximum heart rate ..

The experimental group of resistance training will carry out the training with 8 years of training session with 12 reps with that load will vary according to the 1 RM test.

The composition of the training session is 10 minutes of heating and stretching, 40 minutes of cardiovascular training and 10 minutes of cooling.

ELIGIBILITY:
Inclusion Criteria:

* (American College of Rheumatology). It is necessary to have the presence of room between the elevens criteria for diagnosis:

  * malar erythema
  * discoid lesions
  * photosensitivity
  * oral or nasal ulcers
  * arthritis
  * serositis
  * renal
  * neurological
  * hematological
  * immunological changes
  * antinuclear antibodies.

Exclusion Criteria:

* Patients with hemoglobin level 10gm/dL, sequelae of cardiovascular events, - Respiratory diseases (pulmonary hypertension, pulmonary fibrosis
* Bronchitis, asthma, emphysema)
* Heart failure (NYHA> II)
* History of myocardial ischemia or heart
* Blood pressure> 100 mm Hg.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2009-11; Study Completion 2010-03

PRIMARY OUTCOMES:
Life quality | 12 weeks

SECONDARY OUTCOMES:
Pain | 12 weeks
Strength | 12 weeks
Electromyography | 12 weeks
Aerobic capacity | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo I Abrahão, Principal Investigator — University Federal of São Paulo
Locations (1):
- AmbulatoAmbulatory Specialty Interlagos - General Hospital Grajaú - Association Congregation Santa Catarina, São Paulo, São Paulo, Brazil